CLINICAL TRIAL: NCT02158091
Title: A Phase 1b/2 Study of IPI-145 in Combination With Fludarabine, Cyclophosphamide, and Rituximab (iFCR) in Previously Untreated, Younger Patients With Chronic Lymphocytic Leukemia.
Brief Title: A Phase 1b/2 Study of IPI-145 Plus FCR in Previously Untreated, Younger Patients With CLL
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Secura Bio, Inc. (Industry)
Responsible Party: Principal Investigator, Matthew S. Davids, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-193
Record Dates: First submitted 2014-06-04; First posted 2014-06-06 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — duvelisib; fludarabine; fludarabine phosphate; Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IPI-145 (Experimental): Phase I-Dose escalation will occur using a standard 3-3 dose escalation beginning in dose level 1 with dose cohorts and escalation.
  * Each treatment cycle lasts 28 days (except cycle 1, which is 35 days) during which time IPI-145 will be taken twice daily. The study begins with 1 week of IPI-145 monotherapy.
  * Fludarabine, cyclophosphamide, rituximab (iFCR) - FCR will subsequently be introduced after 1 week and administered at standard dosing for up to 6 cycles, with dose reductions permitted. IPI-145 will be continued through the course of chemotherapy and for up to 2 years maintenance after completing chemotherapy Phase II - 20 additional patients treated with IPI-145 at the Recommended Phase II Dose (RP2D) + fludarabine, cyclophosphamide, rituximab (FCR) with standard dosing.
  Interventions: Drug: IPI-145; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Rituximab

INTERVENTIONS:
Drug: IPI-145 — oral PI3K delta/gamma inhibitor
Drug: Fludarabine — intravenous chemotherapy
  Other Names: Fludara
Drug: Cyclophosphamide — intravenous chemotherapy
  Other Names: Cytoxan®; Neosar®
Drug: Rituximab — intravenous immunotherapy
  Other Names: Rituxan

SUMMARY:
This research study is evaluating a new drug called IPI-145 in combination with the standard drugs fludarabine, cyclophosphamide, and rituximab (FCR), as a possible treatment for chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
Patients who fulfill eligibility criteria will be entered into the trial to receive IPI-145 in combination with the standard drugs fludarabine, cyclophosphamide, and rituximab (FCR). After the screening procedures confirm participation in the research study:

Phase I

The investigators are looking for the highest dose of the combination of study drugs that can be administered safely without severe or unmanageable side effects in participants that have CLL. Not everyone who participates in this research study will receive the same dose of the study drug. The dose given will depend on the number of participants who have been enrolled in the study prior and how well the dose was tolerated.

Phase II:

Patients treated with IPI-145 at the Recommended Phase II Dose (RP2D) + fludarabine, cyclophosphamide, rituximab (FCR) with standard dosing.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of CLL and an indication for treatment as per IW-CLL 2008 criteria
* no prior therapy for CLL
* age 18-65 -- ECOG performance status ≤1

Exclusion Criteria:

* May not be receiving any other study agents
* Known CNS involvement
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because IPI-145 has the potential for teratogenic or abortifacient effects.
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. disease-free for at least 5 years and deemed to be at low risk for recurrence. Individuals with the following cancers are eligible if diagnosed and treated with curative intent within the past 5 years: cervical cancer in situ, localized prostate cancer, and basal cell or squamous cell carcinoma of the skin
* HIV-positive individuals, because of the potential for pharmacokinetic interactions with IPI-145
* Inadequate hepatic function defined by aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 x upper limit of normal (ULN); direct bilirubin >1.5 x ULN, unless due to hemolysis or Gilbert's syndrome
* Inadequate renal function defined by serum creatinine >1.5 x ULN.
* Baseline QTcF >480 ms. NOTE: This criterion does not apply to patients with a left bundle branch block
* Concurrent treatment with any agent known to prolong the QTc interval
* Patients with a history of active tuberculosis within the preceding two years.
* Patients who have had a venous thromboembolic event (e.g., PE/DVT) requiring anticoagulation and who meet any of the following criteria:
* Have been on a stable dose of anticoagulation for <1 month
* Have had a Grade 2, 3 or 4 hemorrhage in the last 30 days
* Are experiencing continued symptoms from their event
* History of alcohol abuse, chronic hepatitis, or other chronic liver disease (other than direct CLL liver involvement)
* Foods or medications that are strong or moderate inhibitors or inducers of CYP3A taken within 1 week prior to study treatment and for the duration of the study
* Unable to receive prophylactic treatment for pneumocystis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-06-27 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2026-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Davids, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Isreal Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in the Phase I portion of the study enrolled in outpatient clinic setting from 6/27/2014 to 1/13/2015 and to the Phase II study from 4/14/2015 to 8/15/2016
Groups:
- Phase I Cohort 1: IPI-145 25mg Once Daily + FCR: Phase I Cohort 1 patients received oral agent IPI-145 25mg daily on days 1-28 of a 28 day cycle, except for Cycle 1, which lasts 35 with a 7 day IPI-145 run in, then will continue daily dosing for 6 cycles and up to 2 years of maintenance. Fludarabine, cyclophosphamide, rituximab (FCR) swill be given standard dosing intravenously (IV) Days 1-3 during week 1 of a cycle for up to 6 cycles, with dose reductions permitted. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
- Phase I Cohort 2 (MTD): IPI-145 25mg Twice Daily + FCR: Phase I Cohort 2 patients received oral agent IPI-145 25mg twice daily ( BID)on days 1-28 of a 28 day cycle, except for Cycle 1, which lasts 35 with a 7 day IPI-145 run in, then will continue daily dosing for 6 cycles and up to 2 years of maintenance. Fludarabine, cyclophosphamide, rituximab (FCR) swill be given standard dosing intravenously (IV) Days 1-3 during week 1 of a cycle for up to 6 cycles, with dose reductions permitted. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
- Phase II Dose Expansion(RP2D)-IPI-145 25mg Twice Daily + FCR: Phase II (MTD)CLL participants received the regimen established in the Phase I study ( January 2015). Phase II Participants received oral IPI-145 25mg twice daily (BID) for up to 6 cycles of combination therapy and 2 years of maintenance ( monotherapy) and received standard dosing if Fludarabine, Cyclophosphamide, and Rituxan (FCR) on days 1-3 of each cycle for up to 6 cycles. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
Period: Overall Study
Arm/Group | Phase I Cohort 1: IPI-145 25mg Once Daily + FCR | Phase I Cohort 2 (MTD): IPI-145 25mg Twice Daily + FCR | Phase II Dose Expansion(RP2D)-IPI-145 25mg Twice Daily + FCR
Started | 6 | 6 | 20
Completed | 4 | 5 | 20
Not Completed | 2 | 1 | 0
Not completed — DLT | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I Cohort 2: IPI-145 25mg Once Daily: Phase I Cohort 2 patients received oral agent IPI-145 25mg twice BID) daily on days 1-28 of a 28 day cycle, except for Cycle 1, which lasts 35 with a 7 day IPI-145 run in, then will continue daily dosing for 6 cycles and up to 2 years of maintenance. Fludarabine, cyclophosphamide, rituximab (FCR) swill be given standard dosing intravenously (IV) Days 1-3 during week 1 of a cycle for up to 6 cycles, with dose reductions permitted. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
- Phase II Dose Expansion ( MTD): IPI 145 25mg BID: Phase II (MTD) CLL participants received the regimen established in the Phase I study ( January 2015). Phase II Participants received oral IPI-145 25mg twice daily (BID) for up to 6 cycles of combination therapy and 2 years of maintenance ( monotherapy) and received standard dosing if Fludarabine, Cyclophosphamide, and Rituxan (FCR) on days 1-3 of each cycle for up to 6 cycles. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
- Total: Total of all reporting groups
Arm/Group | Phase I Cohort 1: IPI-145 25mg Once Daily + FCR | Phase I Cohort 2: IPI-145 25mg Once Daily | Phase II Dose Expansion ( MTD): IPI 145 25mg BID | Total
Number analyzed (Participants) | 6 | 6 | 20 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 20 | 31
  >=65 years | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 6 | 10
  Male | 5 | 3 | 14 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 6 | 5 | 17 | 28
  Unknown or Not Reported | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 6 | 18 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 20 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experienced a Dose Limiting Toxicity (DLT) During Phase I
Description: To assess the safety of IPI145 in combination with FCR in previously untreated younger patients with CLL. DLT is based on the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. DLT refers to toxicities experienced at any time during the study treatment, defined as Grade 3 or greater hematologic toxicity (except Grade 3 or Grade 4 neutropenia or thrombocytopenia that lasts less than or equal to 10 days off treatment), any Grade 3 or greater non-hematologic toxicity (except Grade 3 or greater nausea, vomiting, diarrhea, Grade 3 infusion reactions), Grade 3 asymptomatic laboratory abnormalities that improve to grade 2 or less within 3 days, Inability to receive day 1 therapy of Cycle 2 even after a three week treatment delay due to drug related toxicity from prior cycle, and any Grade 4 or greater elevation in AST ALT values
Time Frame: . Participants were assessed every week or more often as needed during Cycle 1, and every Day 1 Cycles 2 and onward-Dose-limiting toxicities (DLTs) occurring during the first cycle of treatment will be used in determining the Phase II MTD/RP2D
Population: Patients who have received no prior therapy for CLL but who meet IW-CLL 2008 Criteria for requiring treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Cohort 1: IPI-145 25mg Once Daily + FCR | Phase I Cohort 2 (MTD): IPI-145 25mg Twice Daily + FCR
Number analyzed (Participants) | 6 | 6
Participants | 2 | 1

2. Primary Outcome: Number of Patients Who Had a Minimal Residual Disease (MRD) Negative Complete Response (CR) 2 Months After Chemotherapy
Description: To determine the rate of minimal residual disease negative complete response (MRD negative CR) in the bone marrow at 2 months post last cycle of FCR, participants will have a bone marrow biopsy procedure 2 months after completing combination therapy (IPI-145+ FCR) in tandem with a chest,neck, abdomen and pelvic PET CT scan. A central read of the PET CT scan will confirm a radiographic complete response, and the bone marrow pathology and morphology assessments will confirm morphological CR in the bone marrow, while MRD testing will be done by four-color flow cytometry on the bone marrow aspirate with a detection level of 10-4. This will include all patients treated and evaluable at maximum tolerated dose, and at the recommended phase II dose ( RP2D)
Time Frame: 2 months after completion of combination therapy of IPI-145 and FCR
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Phase I MTD and Phase II RP2D: IPI 145 25 mg BID + FCR: Phase I Cohort 2 (MTD) patients and Dose Expansion patients (RP2D) received oral agent IPI-145 25mg twice daily (BID)on days 1-28 of a 28 day cycle, except for Cycle 1, which lasts 35 with a 7 day IPI-145 run in, then will continue daily dosing for 6 cycles and up to 2 years of maintenance. Fludarabine, cyclophosphamide, rituximab (FCR) swill be given standard dosing intravenously (IV) Days 1-3 during week 1 of a cycle for up to 6 cycles, with dose reductions permitted. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
Arm/Group | Phase I MTD and Phase II RP2D: IPI 145 25 mg BID + FCR
Number analyzed (Participants) | 26
Percentage of participants | 23 [9 to 44]

3. Secondary Outcome: Overall Response Rate
Description: Response and progression will be evaluated in this study using the 2008 IW-CLL criteria for CLL (Hallek et al., 2008)
Time Frame: At baseline, End of Cycle 3, and 2 months post FCR
Reporting Status: Not Posted

4. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Toxicity assessments will be done using the CTEP Version 4.0 of the NCI Common Terminology Criteria for Adverse Events (CTCAE) and will include all participants who have received at least 1 dose of IPI-145. Toxicities will be assessed at minimum every week during cycle 1, on Day 1 of every cycle during Cycle 2 onward, and every other cycle Day 1 during maintenance.
Time Frame: Up to 210 days
Reporting Status: Not Posted

5. Secondary Outcome: Rate of Minimal Residual Disease (MRD) in the Peripheral Blood
Description: Participants will have MRD testing in the peripheral blood by four-color flow cytometry at the end of cycle 3, 2 months post combination therapy, and every 6 months thereafter for the duration of treatment and subsequent follow up
Time Frame: 2 Years
Reporting Status: Not Posted

6. Secondary Outcome: Rate of Treatment Related Adverse Effects
Description: Participants will be evaluable for this endpoint if they have had at least 1 dose of study treatment. Toxicities will be assessed at minimum each week during cycle 1, and each day 1 during combination therapy, and then every two months thereafter. CTCAE version 4.0 will be used to assess toxicity term and grading.
Time Frame: 210 days
Reporting Status: Not Posted

7. Secondary Outcome: Determine the Association of Established CLL Prognostic Factors With Clinical Response
Description: Fisher's exact test for categorical variables and Wilcoxon's rank sum test will be used-
Time Frame: 2 Years
Reporting Status: Not Posted

8. Secondary Outcome: Rate of Complete Response and Partial Response
Description: Response and progression will be evaluated in this study using the 2008 IW-CLL criteria for CLL (Hallek et al., 2008)
Time Frame: At baseline, End of Cycle 3, and 2 months post FCR and then per investigator discretion thereafter
Reporting Status: Not Posted

9. Secondary Outcome: Rate of Progression Free Survival
Description: 2008 IW-CLL criteria
Time Frame: At baseline, End of Cycle 3, and 2 months post FCR and then per investigator discretion thereafter
Reporting Status: Not Posted

10. Secondary Outcome: Event Free Survival Rate
Description: Response and progression will be evaluated in this study using the 2008 IW-CLL criteria for CLL (Hallek et al., 2008)
Time Frame: At baseline, End of Cycle 3, and 2 months post FCR and then per investigator discretion thereafter
Reporting Status: Not Posted

11. Secondary Outcome: Duration of Remission Rate
Description: Response and progression will be evaluated in this study using the 2008 IW-CLL criteria for CLL (Hallek et al., 2008)Frequency of follow up visits and scans are per MD discretion. Recommended follow up visits for a minimum of one year
Time Frame: At baseline, End of Cycle 3, and 2 months post FCR and then per investigator discretion thereafter
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events are assessed at minimum every week during cycle 1, and day 1 of every cycle thereafter during combination, and every two cycles thereafter while in maintenance. Treatment duration in cycles was a a median of 6 cycles in Phase I Cohort 1, 4.5 cycles in Phase I Cohort 2 and 5.5 cycles in the Phase II MTD
Description: Maximum grade toxicity by type-Serious AEs were defined as per DFCI criteria: Any grade 2 or 3 unexpected and treatment related event, and all grade 4 and 5 events regardless of attribution to study treatment, and includes events deemed medically important by overall PI. Other AEs were defined as events with the attribution of at least possibly related to the study treatment that did not meet the SAE criteria. CTCAE 4.0 was used in investigator assessment and lab value review.
Groups:
- Phase 1 Cohort 1: IPI-145 25mg Once Daily + FCR: Phase I Cohort 1 patients received oral agent IPI-145 25mg daily on days 1-28 of a 28 day cycle, except for Cycle 1, which lasts 35 with a 7 day IPI-145 run in, then will continue daily dosing for 6 cycles and up to 2 years of maintenance. Fludarabine, cyclophosphamide, rituximab (FCR) swill be given standard dosing intravenously (IV) Days 1-3 during week 1 of a cycle for up to 6 cycles, with dose reductions permitted. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
- Phase 1 Cohort 2: IPI-145 25mg Twice Daily + FCR: Phase I Cohort 2 patients received oral agent IPI-145 25mg twice daily ( BID)on days 1-28 of a 28 day cycle, except for Cycle 1, which lasts 35 with a 7 day IPI-145 run in, then will continue daily dosing for 6 cycles and up to 2 years of maintenance. Fludarabine, cyclophosphamide, rituximab (FCR) swill be given standard dosing intravenously (IV) Days 1-3 during week 1 of a cycle for up to 6 cycles, with dose reductions permitted. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
- Phase II Dose Expansion(MTD)-IPI-145 25mg Twice Daily + FCR: Phase II (MTD)CLL participants received the regimen established in the Phase I study ( January 2015). Phase II Participants received oral IPI-145 25mg twice daily (BID) for up to 6 cycles of combination therapy and 2 years of maintenance ( monotherapy) and received standard dosing if Fludarabine, Cyclophosphamide, and Rituxan (FCR) on days 1-3 of each cycle for up to 6 cycles. Patients are treated until progression without clinical benefit, toxicity, or withdrawal of consent by the patient, or closure of the trial by the Overall PI or regulatory authorities.
Arm/Group | Phase 1 Cohort 1: IPI-145 25mg Once Daily + FCR | Phase 1 Cohort 2: IPI-145 25mg Twice Daily + FCR | Phase II Dose Expansion(MTD)-IPI-145 25mg Twice Daily + FCR
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/20
Serious Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 20/20
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Cohort 1: IPI-145 25mg Once Daily + FCR (N=6) | Phase 1 Cohort 2: IPI-145 25mg Twice Daily + FCR (N=6) | Phase II Dose Expansion(MTD)-IPI-145 25mg Twice Daily + FCR (N=20)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 2 (2)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Investigations) | 1 (1) | 3 (3) | 5 (5)
Leukopenia (Investigations) | 3 (3) | 3 (3) | 4 (4)
Neutrophil Count Decrease (Investigations) | 5 (5) | 4 (4) | 10 (10)
Lymphopenia (Investigations) | 5 (5) | 4 (4) | 5 (5)
Lipase Increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 3 (3)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Drug Induced Liver Injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Inflammatory Bursitis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neck Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Amylase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Pityriasis Rubra Pilaris Reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Cohort 1: IPI-145 25mg Once Daily + FCR (N=6) | Phase 1 Cohort 2: IPI-145 25mg Twice Daily + FCR (N=6) | Phase II Dose Expansion(MTD)-IPI-145 25mg Twice Daily + FCR (N=20)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 3
Alanine aminotransferase increased (Investigations) | 2 | 1 | 8
Alkaline phosphatase increased (Investigations) | 0 | 1 | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 2 | 7
Anorexia (Metabolism and nutrition disorders) | 5 | 3 | 3
Anxiety (Psychiatric disorders) | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 2
Blurred vision (Eye disorders) | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0 | 0
Chills (Vascular disorders) | 4 | 1 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 5 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 4
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 2 | 9
Dizziness (Nervous system disorders) | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 6
Edema limbs (Blood and lymphatic system disorders) | 1 | 1 | 2
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 1
Eye disorders - Other, specify (Eye disorders) | 0 | 2 | 1
Eye pain (Eye disorders) | 1 | 0 | 0
Fatigue (General disorders) | 6 | 6 | 10
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2
Fever (Immune system disorders) | 4 | 4 | 9
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flu like symptoms (Immune system disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4 | 2 | 4
General disorders and administration site conditions - Other, specify (General disorders) | 3 | 0 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Headache (Nervous system disorders) | 3 | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1
Infections and infestations - Other, specify (Infections and infestations) | 2 | 0 | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 3 | 1 | 1
Investigations - Other, specify (Investigations) | 0 | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2
Lipase increased (Investigations) | 0 | 1 | 1
Lung infection (Infections and infestations) | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 3 | 2 | 4
Lymphocyte count increased (Investigations) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 | 4 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 5 | 12
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 5 | 3 | 9
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Pain (General disorders) | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 3
Pharyngeal necrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Platelet count decreased (Investigations) | 6 | 2 | 10
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 1 | 0
Serum amylase increased (Investigations) | 0 | 1 | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 | 2 | 0
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 | 4 | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 1 | 0
Syncope (Nervous system disorders) | 1 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Tooth discoloration (Gastrointestinal disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 3 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1 | 0
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1 | 4
Weight gain (Investigations) | 1 | 0 | 0
Weight loss (Investigations) | 2 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
White blood cell decreased (Investigations) | 6 | 4 | 4
Wound infection (Infections and infestations) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT02158091/Prot_SAP_000.pdf